CLINICAL TRIAL: NCT00491933
Title: Comparison of Quantiferon-TB Gold Assay With Tuberculin Skin Testing in the Assessment of Latent Mycobacterium Tuberculosis Infection in Patients Candidate to Treatment or Treated With TNFα Antagonists
Brief Title: Quantiferon-TB Gold in the Assessment of Latent TB in Patients Candidate to Treatment or Treated With TNFα Antagonists
Acronym: TNFTB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-RHEU-2007-001
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Rheumatoid Arthritis; Spondylarthritis; Tuberculosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Quantiferon-TB Gold assay
Procedure: Tuberculin skin test

SUMMARY:
The purpose of this study is to evaluate the value of Quantiferon-TB Gold (QFT-G) assay in the screening for latent tuberculosis infection (LTBI) in rheumatologic patients due to start or on treatment with TNFα antagonists. The results of QFT-G will be compared to tuberculin skin testing (TST) and correlated to clinical and demographic data. The study hypothesis is that the inclusion of QTF-G in the screening strategy will allow a more accurate assessment of LTBI infection.

DETAILED DESCRIPTION:
Treatment with TNFα antagonists is associated with an increased risk of active tuberculosis. Screening for LTBI and adherence to published guidelines have been shown to greatly decrease the risk of active tuberculosis. However, the best screening strategy is still object of debate. The validity of TST in patients on immunosuppressive treatment has been questioned. Recently, interferon-γ assays based on RD1-specific antigens have shown to cause less confounding by BCG vaccination and from most non-tuberculosis mycobacteria than TST, and have shown improved accuracy over TST in several settings. However, data on their use in rheumatologic patients are limited, and their superiority in patients on immunosuppressive treatment is unclear since indeterminate results may limit their clinical usefulness in this setting.

Purpose of the study is to investigate the added value of the inclusion of QTF-G assay in the screening strategy of LTBI in rheumatologic patients before and during treatment with TNFα antagonists.

The study will compare the results of TST with the results of QFT-G assay in rheumatologic patients being evaluated for treatment with anti-TNFα agents or already on treatment with anti-TNFα agents. The rate of positive and negative results of the two test will be compared, end results correlated to clinical and demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatological diseases being evaluated for treatment with TNFα antagonists or on treated with TNFα antagonists

Exclusion Criteria:

* Unable to sign informed consent
* Known hypersensitivity to tuberculin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Concordance between the QFT-G assay and the tuberculin skin test
Correlation of the test results to the patient's risk of LTBI

SECONDARY OUTCOMES:
Factors associated with discordance between the TST and the QFT-G test
Frequency of indeterminate results

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antivalle, MD, Principal Investigator — Ospedale L. Sacco - Polo Universitario, Milano, Italy
Locations (1):
- Rheumatology Unit, Ospedale L. Sacco Polo Universitario, Milan, Italy

REFERENCES:
- [Background] Gomez-Reino JJ, Carmona L, Valverde VR, Mola EM, Montero MD; BIOBADASER Group. Treatment of rheumatoid arthritis with tumor necrosis factor inhibitors may predispose to significant increase in tuberculosis risk: a multicenter active-surveillance report. Arthritis Rheum. 2003 Aug;48(8):2122-7. doi: 10.1002/art.11137. PMID 12905464
- [Background] British Thoracic Society Standards of Care Committee. BTS recommendations for assessing risk and for managing Mycobacterium tuberculosis infection and disease in patients due to start anti-TNF-alpha treatment. Thorax. 2005 Oct;60(10):800-5. doi: 10.1136/thx.2005.046797. Epub 2005 Jul 29. PMID 16055611
- [Background] Ferrara G, Losi M, Meacci M, Meccugni B, Piro R, Roversi P, Bergamini BM, D'Amico R, Marchegiano P, Rumpianesi F, Fabbri LM, Richeldi L. Routine hospital use of a new commercial whole blood interferon-gamma assay for the diagnosis of tuberculosis infection. Am J Respir Crit Care Med. 2005 Sep 1;172(5):631-5. doi: 10.1164/rccm.200502-196OC. Epub 2005 Jun 16. PMID 15961696